CLINICAL TRIAL: NCT01305304
Title: Magnetic Resonance Technique in the Assessment of Exercise-induced Long- and Short-Term Changes in Cardiac Function and Morphology
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Federal Office of Sports, Switzerland (Other Government)
Responsible Party: Dr.phil.nat. Dr.sci.med. Michael Ith, Dept. of Diagnostic, Interventional and Pediatric Radiology (DIPR) University & Inselspital Bern
Other Study IDs: KEK 005/010 B
Record Dates: First submitted 2011-02-11; First posted 2011-02-28 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Myocardial Ischemia; Myocardial Infarction; Ventricular Remodeling; Myocardial Contraction; Ventricular Hypertrophy
MeSH Terms: conditions — Myocardial Ischemia; Myocardial Infarction; Ventricular Remodeling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 15 healthy male "veteran" runners (marathon, triathlon, orienteering) aged between 40 and 65 years with a history of competitive running at a national level during a period of at least 5 years, implicating normally a runner career with at least 50km per week over more than 10 years
  Interventions: Other: repeated long term endurance exercise
- 2: 15 healthy male volunteers, matched for age and bmi, without a history of competitive physical exercise (i.e. sedentary controls)
  Interventions: Other: Other

INTERVENTIONS:
Other: repeated long term endurance exercise — competitive running at a national level during a period of at least 5 years (i.e. approximately 50km per week over more than 10 years)
  Groups: 1
Other: Other — No history of endurance sports activity
  Groups: 2

SUMMARY:
Until now it has been assumed that regular endurance training has a positive influence on cardiac function and that the positive effect increases with increasing intensity. However, little is known about the effects of intense endurance stress on the heart. According to current knowledge repeated exposure to strenuous endurance activity may lead to minor but possibly irreversible damage to the heart with resultant scarring of the heart's muscle.

Within this study the investigators attempt to find out by different analytical methods - in particular magnetic resonance imaging (MRI) and ultrasound of the heart - to what extent the heart muscle is affected by long term intense endurance exercise and which changes in cardiac function and morphology can possibly be found. Therefore the investigators compare former national competitive endurance athletes with sedentary controls.

DETAILED DESCRIPTION:
Background

Despite the well documented cardio-protective effects of aerobic exercise of moderate intensity, short- and long-term consequences of strenuous exercise are less clear. There is increasing evidence that maintaining a high cardiac workload over a prolonged duration may result in transient impairment of cardiac function. Recent studies have also reported a transient increase in cardiac biomarkers after prolonged strenuous exercise. While in patients with cardiac disease the presence of cardiac dysfunction and increased cardiac biomarkers generally reflects myocardial damage, the impact of these observations in athletes is ill defined. It is a matter of concern whether in athletes such findings simply reflect a reversible response or whether repetitive events may lead to an accumulative cardiac damage. Traditional echocardiographic methods used to determine potential cardiac changes in morphology or function are investigator-dependent and may be subject to interference by cardiac pre- and afterload. Cardiac magnetic resonance imaging provides an investigator-independent and objective method to quantify cardiac dimensions and function. Delayed contrast enhancement MR imaging is a highly reproducible cardiovascular magnetic resonance imaging technique to directly visualize myocardial edema, necrosis and fibrosis.

Objective

To use cardiac and delayed contrast enhancement magnetic resonance imaging in combination with echocardiographic methods to to assess whether athletes involved in prolonged strenuous exercise over years reveal persistent alterations of cardiac morphology and function.

Methods

Cardiac and delayed contrast enhancement magnetic resonance imaging will be used in combination with echocardiographic methods to investigate whether involvement in prolonged strenuous exercise over years leads to changes in cardiac function and morphology. Therefore we study and compare 15 veteran elite athletes and 15 sedentary controls. The use of cardiac MRI and delayed contrast enhancement magnetic resonance imaging techniques will be paralleled by echocardiographic and tissue Doppler measurements to allow comparative analyses of the two methods.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-65y
* Healthy
* history of national competitive endurance running (cases)
* no history of endurance running (controls)

Exclusion Criteria

* Contraindication for MRI
* History of relevant cardiac disease (including cardiomyopathies)
* coronary heart disease
* coronary abnormalities
* cardiovascular risk factors
* History of any chronic disease
* drug abuse
* Arrhythmias which make adequate echocardiography unfeasible (such as atrial fibrillation or bundle-branch blocks)

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: residents of Switzerland, either with history of national competitive endurance running (cases) or without history of endurance running (controls)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
cardiac fibrosis (area in cm^2) on late contrast enhanced MR images | at subject enrollment (cross-sectional design)

SECONDARY OUTCOMES:
systolic/diastolic function and contractility measured by echocardiography | at subject enrollment (cross-sectional design)
various parameters of cardiac function and morphology assessed with MRI and echocardiography | at subject enrollment (cross-sectional design)
anthropometric data | at subject enrollment (cross-sectional design)
VO2max | at subject enrollment (cross-sectional design)
resting-ECG | at subject enrollment (cross-sectional design)
stress-ECG | at subject enrollment (cross-sectional design)
blood analyses | at subject enrollment (cross-sectional design)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ith, PhD, PhD/MD, Principal Investigator — Dept. of Diagnostic, Interventional and Pediatric Radiology, University Hospital Bern; Christoph Stettler, MD, Principal Investigator — Division of Endocrinology, Diabetes and Clinical Nutrition, University Hospital Bern
Locations (1):
- Dept. of Diagnostic, Interventional and Pediatric Radiology, University Hospital Bern, Bern, Switzerland